CLINICAL TRIAL: NCT01891331
Title: A Phase 2A, Randomized, Double-Blind, Dose Ranging Study to Evaluate the Efficacy and Safety of VT-1161 Oral Tablets Compared to Fluconazole in the Treatment of Patients With Moderate to Severe Acute Vulvovaginal Candidiasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral VT-1161 in Patients With Acute Vaginal Candidiasis (Yeast Infection)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viamet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-004
Record Dates: First submitted 2013-06-17; First posted 2013-07-03 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Candidiasis, Vulvovaginal
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- VT-1161 300mg QD (Experimental)
  Interventions: Drug: VT-1161
- VT-1161 600mg QD (Experimental)
  Interventions: Drug: VT-1161
- VT-1161 600mg BID (Experimental)
  Interventions: Drug: VT-1161
- Fluconazole 150mg (Active Comparator)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: VT-1161
  Arms: VT-1161 300mg QD; VT-1161 600mg BID; VT-1161 600mg QD
Drug: Fluconazole
  Arms: Fluconazole 150mg

SUMMARY:
The purpose of this study is to determine if the novel oral agent VT-1161 is safe and effective in treating patients with acute vulvovaginal candidiasis (also referred to as yeast infection). VT-1161 has been designed to inhibit CYP51, an enzyme essential for fungal growth. Inhibition of CYP51 results in the accumulation of chemicals know to be toxic to the fungus. CYP51 is the molecular target of the class of drugs referred to as 'azole antifungals'. All currently approved azole drugs have poor selectivity for CYP51 and this results in many of the side effects associated with the azole antifungals. The safety profile of the class similarly limits use in chronic treatment of non-life-threatening fungal infections. VT-1161 has been design to be safer and more active against the fungal species typically responsible for vaginal yeast infections (i.e. vulvovaginal candidiasis).

ELIGIBILITY:
Key Inclusion Criteria:

* Females ≥18 and <65 years
* Clinical diagnosis of symptomatic acute VVC
* Positive KOH .At least one vulvovaginal sign (vulvovaginal erythema, edema, or excoriation).
* At least one vulvovaginal symptom (vulvovaginal itching, burning, or irritation)
* A minimum composite vulvovaginal signs and symptoms score of ≥6
* must be be able to swallow capsules

Exclusion Criteria:

* Evidence of major organ system disease
* History of cervical cancer
* History of diabetes mellitus
* Pregnant
* Recent use of systemic antifungal drugs or systemic antimicrobial therapy for any reason
* Recent use of drugs to treat vaginal infections
* Recent use of immunosuppressive therapies

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Altus Research, Lake Worth, Florida
  - Healthcare Clinical Data, Inc, North Miami, Florida
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Lyndhurst Clinical Research, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Drexel Vaginitis Center, Philadelphia, Pennsylvania
  - Brownstone Clinical Trials, LLC, Irving, Texas
  - Harborview ID Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Vanreppelen G, Nysten J, Baldewijns S, Sillen M, Donders G, Van Dijck P. Oteseconazole (VIVOJA) for prevention of recurrent vulvovaginal candidiasis. Trends Pharmacol Sci. 2023 Jan;44(1):64-65. doi: 10.1016/j.tips.2022.10.004. Epub 2022 Nov 14. No abstract available. PMID 36396498
- [Derived] Brand SR, Sobel JD, Nyirjesy P, Ghannoum MA, Schotzinger RJ, Degenhardt TP. A Randomized Phase 2 Study of VT-1161 for the Treatment of Acute Vulvovaginal Candidiasis. Clin Infect Dis. 2021 Oct 5;73(7):e1518-e1524. doi: 10.1093/cid/ciaa1204. PMID 32818963

RESULTS

PARTICIPANT FLOW:
Groups:
- VT-1161 300mg QD: VT-1161 300mg once daily for 3 days
- VT-1161 600mg QD: VT-1161 600mg once daily for 3 days
- VT-1161 600mg BID: VT-1161 600mg twice daily for 3 days
- Fluconazole 150mg: Single dose of fluconazole 150mg
Period: Overall Study
Arm/Group | VT-1161 300mg QD | VT-1161 600mg QD | VT-1161 600mg BID | Fluconazole 150mg
Started | 14 | 12 | 14 | 15
Completed | 12 | 10 | 13 | 13
Not Completed | 2 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VT-1161 300mg QD | VT-1161 600mg QD | VT-1161 600mg BID | Fluconazole 150mg | Total
Number analyzed (Participants) | 14 | 12 | 14 | 15 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (12.01) | 38.2 (11.77) | 27.6 (7.37) | 31.3 (8.22) | 32.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 14 | 15 | 55
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Therapeutic Cure at 28 Days for All-Analysis Population
Description: For this trial, therapeutic cure was defined as mycological AND clinical cure. Mycological cure was defined as a negative fungal culture for Candida species. Clinical cure was defined as all of the following:
  1. complete resolution of signs and symptoms pertaining to vulvovaginal candidiasis;
  2. any new sign or symptom observed at 28 days determined by investigator to not be related to vulvovaginal candidiasis;
  3. no use of any other antifungal drug therapy for treatment of vulvovaginal irritation and/or pruritus by subject.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VT-1161 300mg QD | VT-1161 600mg QD | VT-1161 600mg BID | Fluconazole 150mg
Number analyzed (Participants) | 14 | 12 | 14 | 15
Participants | 9 | 9 | 11 | 10

ADVERSE EVENTS:
Arm/Group | VT-1161 300mg QD | VT-1161 600mg QD | VT-1161 600mg BID | Fluconazole 150mg
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 10/14 | 6/12 | 3/14 | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VT-1161 300mg QD (N=14) | VT-1161 600mg QD (N=12) | VT-1161 600mg BID (N=14) | Fluconazole 150mg (N=15)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Conjunctivitis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 2
Esophageal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitits (Infections and infestations) | 1 | 0 | 0 | 0
Trichamoniasis (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Vaginitis Bacterial (Infections and infestations) | 2 | 1 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Urine Odor Abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine Hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither institution nor principal investigator shall publish the results of the trial without prior written consent of the sponsor, which it may withhold in its sole discretion.